CLINICAL TRIAL: NCT01037049
Title: Is Greater Downstaging and Tumour Regression Observed When Surgery is Delayed to 12 Weeks After Completion of Chemoradiotherapy vs 6 Weeks?
Brief Title: Optimum Timing for Surgery After Pre-operative Radiotherapy 6 vs 12 Weeks
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CCR3227
Record Dates: First submitted 2009-12-18; First posted 2009-12-21 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Adenocarcinoma of the Rectum; Adenocarcinoma; Adenocarcinoma, Mucinous; Carcinoma; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neoplasms; Neoplasms, Cystic, Mucinous, and Serous; Colorectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Digestive System Diseases; Gastrointestinal Diseases; Intestinal Diseases; Rectal Diseases
Keywords: Rectal Cancer; 6vs12; 6 vs 12; Cancer; CRM; Circumferential Resection Margin; Quality of Life; MRI; Radiology; Abdominoperineal Excision; Anterior Resection; Surgery; Pathology; Radiotherapy
MeSH Terms: conditions — Rectal Neoplasms; Adenocarcinoma; Adenocarcinoma, Mucinous; Carcinoma; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neoplasms; Neoplasms, Cystic, Mucinous, and Serous; Colorectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Digestive System Diseases; Gastrointestinal Diseases; Intestinal Diseases; Rectal Diseases | interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (No Intervention): Patients who have surgery at 6 weeks after radiotherapy/chemoradiotherapy
- Group 2 (Experimental): Patients who have surgery at 12 weeks after radiotherapy/chemoradiotherapy
  Interventions: Other: Patients who have surgery at 12 weeks after radiotherapy/chemoradiotherapy

INTERVENTIONS:
Other: Patients who have surgery at 12 weeks after radiotherapy/chemoradiotherapy
  Arms: Group 2

SUMMARY:
The aim of this study is to determine whether greater rectal cancer downstaging and regression occurs when surgery is delayed to 12 weeks after completion of radiotherapy/chemotherapy compared to 6 weeks.

Hypothesis: Greater downstaging and tumour regression is observed when surgery is delayed to 12 weeks after completion of CRT compared to 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Aged > 18
* Informed written consent
* Histological confirmation of adenocarcinoma of rectum
* Undergoing pre-operative radiotherapy/ chemotherapy
* Completion of pre-operative treatment

Exclusion Criteria:

* Aged < 18
* Absence of pre-operative RT/CT
* Medical/ psychiatric conditions that compromise the patients ability to give informed consent
* Contra-indications to MRI, i.e. hip prothesis, cardiac pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2009-10-16 (Actual); Primary Completion 2014-12-08 (Actual); Study Completion 2019-12-08 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be the difference in the proportion of patients in each arm, downstaged according to T stage [on MRI]. | 6-12 weeks

SECONDARY OUTCOMES:
Tumour response using SUV measurements [PET/CT], N downstaging and Tumour Regression Grade downstaging [on MRI]. | 3 months
Difference in proportion of patients in each arm undergoing sphincter saving surgery. | 3 months
Morbidity, 30 day mortality and CRM (circumferential resection margin) positivity. | 3 months
An analysis will also be undertaken using multivariate and linear regression analysis to evaluate the association of ypT and ypN stage as a potential independent predictors of SUV (max) baseline and after radiotherapy (pre-surgery) in the two arms. | 3 months
Local and distant recurrence rates. | 5 years
Radiotherapy related toxicity rates. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Diana Tait, Principal Investigator — Royal Marsden NHS Foundation Trust; Gina Brown, Principal Investigator — Royal Marsden Hospitals NHS Foundation Trust
Locations (23):
- Hospital Alemão Oswaldo Cruz, São Paulo, Brazil
- Jewish General Hospital, Montreal, Quebec, Canada
- Bank of Cyprus Oncology Centre, Nicosia, Cyprus
- United Kingdom (20):
  - Hinchingbrooke Hospital, Huntingdon, Cambridgeshire
  - County Durham and Darlington NHS Trust (University Hospital of North Durham), Durham, County Durham
  - North Tees and Hartlepool NHS Trust (University Hospital of North Tees), Stockton-on-Tees, County Durham
  - Dorset County Hospital NHS Foundation Trust, Dorchester, Dorset
  - Poole Hospital NHS Foundation Trust, Poole, Dorset
  - Essex County Hospital, Colchester, Essex
  - Portsmouth Hospitals NHS Trust (Queen Alexandra Hospital), Portsmouth, Hampshire
  - Medway NHS Foundation Trust, Gillingham, Kent
  - North West London Hospitals NHS Trust (Northwick Park Hospital), Harrow, Middlesex
  - James Paget University Hospitals NHS Foundation Trust, Great Yarmouth, Norfolk
  - Epsom and St Helier's Hospitals NHS Trust, Carshalton, Surrey
  - St Richard's Hospital, Chichester, West Sussex
  - Mid Yorkshire Hospitals NHS Trust (Pinderfields Hospital), Wakefield, West Yorkshire
  - Royal United Hospital NHS Trust, Bath
  - Sandwell and West Birmingham Hospitals NHS Trust, Birmingham
  - Croydon University Hospital, Croydon
  - St Bartholomew's Hospital, London
  - St George's Healthcare NHS Trust, London
  - Pennine Acute Hospitals NHS Trust, Manchester
  - Royal Marsden NHS Trust, Sutton